CLINICAL TRIAL: NCT05163262
Title: Descriptive and Prospective Study of Sphincter Disorders in the Severe Traumatic Brain Injury Population
Acronym: TCG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of staff to carry out the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP211155
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Sexuality; Sexual disorders; bladder-sphincter dysfunctions; anorectal disorders
MeSH Terms: conditions — Brain Injuries, Traumatic; Sexuality; Sexual Dysfunction, Physiological; Rectal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Addition of a sexuality questionnaire during patient follow-up within 3 months after inclusion, 6 months after and at one year
  Interventions: Other: sexuality questionnaire

INTERVENTIONS:
Other: sexuality questionnaire — Questionnaire evaluating the sexuality of head trauma victims by comparing their sexual focus, the quality of their relationship, their self-esteem, their mood before the trauma to their current situation

SUMMARY:
Severe traumatic brain injury (TCI), defined by an initial GCS of ≤ 8 and/or admitted to a neurosurgical intensive care unit, are responsible for diffuse brain lesions that can lead to multiple deficits, including impairment of sphincter functions: bladder, rectal and sexual.

Bladder-sphincter disorders are very common after a TBI. Urinary incontinence predominates, with a prevalence varying from 50 to 100% in the acute period following a TBI.

The variability of the clinical data is explained by the heterogeneity of the populations studied (severity of TBI, duration of coma, time to care) and the tools used to objectify sphincter disorders. The interest of this study is to make an evaluation and a prospective follow-up of sphincter disorders in this population during one year.

DETAILED DESCRIPTION:
A first visit, planned as part of the care, within 3 months of TBI with a clinical examination and 8 to 11 questionnaires, depending on your sex and your transit, to assess cognitive functions, the sphincter sphere, the autonomy and mood achieved as part of your usual care. These questionnaires will be taken with the doctor during consultation, As part of the research, patient will be asked to additionally answer the sexuality questionnaire consisting of 23 questions.

The same visit will be carried out at 6 months and at 1 year, also planned as part of the usual care.

If beyond 6 months vesico-sphincter complaints persist, a urodynamic examination will be realised in order to compare subjective complaints with a urodynamic examination (flowmeter, cystomanometry with +/- pressure / flow rate curve, sphincterometry).

This is a single-center research. The patients will be included in the neurosurgical intensive care unit of the Pitié Salpêtrière hospital and will be followed in the Physical Medicine and Rehabilitation unit of the same hospital.

ELIGIBILITY:
Inclusion Criteria:

* Have been the victim of a serious head trauma (initial glasgow ≤ 8 and / or admitted to neurosurgical resuscitation for less than 3 months
* Admitted to Neurosurgical Resuscitation at Pitié-Salpêtrière
* Aged 18 to 70
* Good written and oral comprehension of the French language
* Glasgow score = 15 at the time of inclusion and able to say no to opposition
* Patient information and not opposition

Exclusion Criteria:

* Severe comprehension disorders
* History of vesico-sphincteric disorders before TC
* Neurological and psychiatric history
* Patient not affiliated to a social security scheme or entitled
* Patient under guardianship / curators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through the sexuality questionary | 3 month after inclusion
  Overall score from 15 to 75, threshold 45
  * Sexual functioning (8 questions): score from 8 to 40, threshold 24
  * Quality of Relationship and Self-Esteem (5 questions): score from 5 to 25, threshold 15
  * Mood (2 questions): score from 2 to 10, threshold 6
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through the Female sexual function Index | 3 month after inclusion
  The presence of these disorders will be reported subjectively by patients the lower the score, the more complaints the patient has, there is no pathological threshold.
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through the Premature Ejaculation Profile | 3 month after inclusion
  The presence of these disorders will be reported subjectively by patients the lower the score, the more complaints the patient has, there is no pathological threshold.
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through the abridged IIEF-5 questionary, | 3 month after inclusion
  referred to as the Sexual Health Inventory of Men (SHIM) = SHIM-IIEF 5: Erectile dysfunction severe (score of 5 to 10), moderate (11 to 15), mild (16 to 20), normal erectile function (21 to 25) and not interpretable (1 to 4)
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through the Wexner score if diarrhea | 3 month after inclusion
  the higher the score, the greater the achievement, there is no defined threshold.
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through The Neurogenic Bowel Dysfunction if constipation | 3 month after inclusion
  a score between 0-6 indicates very minimal impairment, 7-9: minimal; 10-13 moderate; ≥ 14 severe
evaluate the prevalence and typology of sphincter disorders in patients presenting a TCG of less than 3 months and admitted to the neurosurgical unit of the Pitié-Salpêtrière through the Urinary Symptom Profile questionary | 3 month after inclusion
  overall score ≥ 5 indicates a bladder complaint

SECONDARY OUTCOMES:
The course of sphincter disorders will occur: • By clinical evaluation | less than 3 months, 6 months and 1 year from TC
The course of sphincter disorders will occur: The subjective complaints will be compared with a urodynamic examination (flowmeter, cystomanometry with +/- pressure / flow rate curve, sphincterometry in order to objectify the disorders if they persist | less than 3 months, 6 months and 1 year from TC
  The urodynamic examination allows if there is a neurological bladder (detrusor hyperactivity, hypocontractility, vesico-sphincteric dyssynergy) to corroborate the patient's complaints and therefore to guide the therapeutic management (anticholinergics, alphablocker, auto- surveys, transcutaneous neurostimulation).
The course of sphincter disorders will occur:By self-administered questionaries less than 3 months, 6 months and 1 year from TC. | less than 3 months, 6 months and 1 year from TC
  The self-questionaries are the same as those for the main criterion allowing the diagnosis of sphincter disorders.
The results of the TBI sexuality questionary will be compared with the reference questionaries that are not specific to head trauma in order to assess the correlation between these questionaries. | less than 3 months, 6 months and 1 year from TC
  in men: ▪ the abridged IIEF-5questionaries, referred to as the Sexual Health Inventory of Men (SHIM) = SHIM-IIEF 5 and Premature Ejaculation Profile (PEP)
  • in women Female sexual function Index (FSFI)
correlate whether the patients who have the most vesicosphincter complaints are the patients with the most more severe and / or the most depressed or vice versa | less than 3 months, 6 months and 1 year from TC
  Tests evaluating cognitive functions (MOCA / BREF), patients' functional recovery (GOSE / MIF) and thymic state (HADS),

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine Physique et Réadaptation , Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No